CLINICAL TRIAL: NCT05803330
Title: Clinical Study of Abandonment of Intravenous Volume Expansion After Preoperative Use of α-blockers in Patients With Adrenal Pheochromocytoma
Brief Title: Study of Alpha-blockers Alone During Preoperative Preparation in Patients With Pheochromocytoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kunwu Yan,MM (Other)
Responsible Party: Sponsor-Investigator, Kunwu Yan,MM, Research Project Leader, Handan First Hospital
Organization: Handan First Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202303-1
Record Dates: First submitted 2023-03-14; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Adrenal Pheochromocytoma; Hemodynamic
MeSH Terms: conditions — Pheochromocytoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PXB combined with venous dilation group (No Intervention): Use of PXB combined with intravenous volume expansion during preoperative preparation in patients with pheochromocytoma
- PXB group (Experimental): PXB alone during preoperative preparation in patients with pheochromocytoma
  Interventions: Drug: Abandonment of intravenous volume expansion during preoperative preparation in patients with pheochromocytoma

INTERVENTIONS:
Drug: Abandonment of intravenous volume expansion during preoperative preparation in patients with pheochromocytoma — Abandonment of intravenous volume expansion with alpha-blockers during preoperative preparation in patients with pheochromocytoma
  Arms: PXB group

SUMMARY:
Study of the relationship between hemodynamic stability and preoperative intravenous rehydration in patients with pheochromocytoma

DETAILED DESCRIPTION:
All patients were subclassified into either the hemodynamic stability group (HS group) or the hemodynamic instability group (HU group) according to whether intraoperative hemodynamic instability occurred. Differences in data between the two groups were examined, and the risk factors for intraoperative hemodynamic instability were analyzed using logistic regression.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of adrenal pheochromocytoma Must be able to swallow tablets

Exclusion Criteria:

Bilateral or multiple pheochromocytomas. Ectopic pheochromocytoma

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
intraoperative mean arterial pressure | During surgery
  an intraoperative mean arterial pressure <60 mmHg is considered to be hemodynamically unstable

CONTACTS AND LOCATIONS:
Overall Officials: kunwu yan, Master, Principal Investigator — Handan First Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meijs AC, Snel M, Corssmit EPM. Pheochromocytoma/paraganglioma crisis: case series from a tertiary referral center for pheochromocytomas and paragangliomas. Hormones (Athens). 2021 Jun;20(2):395-403. doi: 10.1007/s42000-021-00274-6. Epub 2021 Feb 11. PMID 33575936
- [Background] Challis BG, Casey RT, Simpson HL, Gurnell M. Is there an optimal preoperative management strategy for phaeochromocytoma/paraganglioma? Clin Endocrinol (Oxf). 2017 Feb;86(2):163-167. doi: 10.1111/cen.13252. Epub 2016 Oct 24. PMID 27696513
- [Background] Randle RW, Balentine CJ, Pitt SC, Schneider DF, Sippel RS. Selective Versus Non-selective alpha-Blockade Prior to Laparoscopic Adrenalectomy for Pheochromocytoma. Ann Surg Oncol. 2017 Jan;24(1):244-250. doi: 10.1245/s10434-016-5514-7. Epub 2016 Aug 25. PMID 27561909
- [Background] Bihain F, Nomine-Criqui C, Guerci P, Gasman S, Klein M, Brunaud L. Management of Patients with Treatment of Pheochromocytoma: A Critical Appraisal. Cancers (Basel). 2022 Aug 9;14(16):3845. doi: 10.3390/cancers14163845. PMID 36010839